CLINICAL TRIAL: NCT05860231
Title: Comparative Mixed Study of the Foley Catheter With the T-Control® Catheter in Patients With Long-term Catheterization
Brief Title: Comparative Study Between Foley and T-Control® Catheter in Patients With Long-term Catheterization
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to issues with investigational device impacting its functionality and user handling. The sponsor decided to implement necessary design and/or material modifications to improve performance and safety before resuming recruitment.
Sponsor: Rethink Medical SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RM-TCONTROL-2022-02
Record Dates: First submitted 2023-04-24; First posted 2023-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Catheter-Associated Urinary Tract Infection; Catheter Related Complication; Quality of Life
Keywords: Catheterisation; T-Control; Foley catheter; Bladder catheter; Urinary catheter

STUDY DESIGN:
Masking Description: Data analysis will be blinded to the intervention arm as well as the laboratories that will carry out the analysis of the urine and catheter samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Foley catheter) (Active Comparator): When randomly allocated to this arm, a conventional Foley-type catheter will be inserted during all the study period (4 weeks). At day 28 after inclusion, the patient will be called for a follow-up visit to remove the catheter.
  Interventions: Device: Foley catheter
- T-Control arm (Experimental): When randomly allocated to this arm, the T-Control catheter will be inserted during all the study period (4 weeks). At day 28 after inclusion, the patient will be called for a follow-up visit to remove the catheter.
  Interventions: Device: T-Control catheter

INTERVENTIONS:
Device: Foley catheter — Silicone Foley catheters are transurethral balloon catheters used for the treatment of bladder emptying disorders, as well as for drainage of urine from the urinary tract, continuous fluid irrigation, and/or medication administration. Its use is suitable for a prolonged period of no more than 29 days and is used in Urology, Internal Medicine, Surgery, Obstetrics and Gynaecology Services.
  For this study, conventional Foley-type catheters whose use is approved in Spain for routine use will be used. Silicone Foley catheters, usually available in 2- and 3-way, are made of silicone and consist of a body, drainage funnel, inflation funnel, irrigation funnel (if present, only on 3-way catheters) and balloon valve. The product is sterile and single use.
  Arms: Control arm (Foley catheter)
Device: T-Control catheter — The T-control® catheter is a flexible, sterile silicone tube with an inflatable balloon at the distal tip, a polytetrafluroethylene membrane integrated into its body, and a sliding fluid control valve. The valve, built into the catheter, provides additional functions to the catheter, such as turning urine flow on and off after insertion (functions currently provided by accessories such as caps or valves) and controlling urination during the insertion process (function that is not provided by any other device). In this way, accidental loss of urine can be avoided from the first moment of use until its withdrawal. Additionally, it has a safety cap that reduces the possibility of accidental movements of the valve before use or during transport and fixing. The design has been developed in such a way that, once inserted, it facilitates autonomous use even for the elderly or patients with limited manual dexterity. The device is sterile and single use, like any conventional Foley catheter.
  Arms: T-Control arm

SUMMARY:
This is a comparative, randomized, controlled pilot study. The main objective of this study is to evaluate the efficacy, comfort, and patient experience in people with long-term bladder catheterization with T-Control® versus patients with a conventional Foley-type catheter.

DETAILED DESCRIPTION:
This is a mixed study, in which, on the one hand, a pilot, randomized, two-arm comparative study will be carried out to compare the T-Control® catheter versus the Foley-type catheter in patients with long-term catheterization, monitoring the patient from the insertion of the catheter until its removal or change (4 weeks). On the other hand, a study will be carried out with qualitative methodology, through discussion groups to explore the experience of the patients who participated in the part of the study with quantitative methodology.

The sample of patients will be recruited in the urology service of Hospital 12 de Octubre. The identification of patients eligible to participate will be carried out by members of the urology service staff. During the inclusion period, all those patients who require a long-term bladder catheter change will be invited to participate, who will be interviewed at an initial visit, where the inclusion and exclusion criteria will be checked, the patients will receive information about the study, they will decide whether or not they want to participate, they will sign and deliver the written informed consent and they will be randomly included in the study in one of the two arms, study group (patients catheterized with T-Control®) and control group (patients catheterized with conventional Foley). Both inclusion and randomization will be performed by the investigator responsible for catheter insertion. During this initial visit, patients who decide to participate and meet the criteria will receive an incident diary to keep and record follow-up, and the catheter will be inserted.

Four weeks after bladder catheter insertion, patients will be called for a follow-up visit, during which the study catheter will be removed or replaced.

If the patient is selected for the discussion group, during this follow-up visit they will be informed of the date and place where the qualitative study will be carried out. The discussion groups will be moderated by a researcher with experience in this field who does not have a therapeutic relationship with the participants.

ELIGIBILITY:
Inclusion Criteria:

* Man or women equal or over 18 years old
* Patients who require a change of bladder catheter.
* Indication of bladder catheterization for 4 weeks.
* Maintained cognitive and physical capacity for self-monitoring of the T-Control ® catheter valve.
* Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Symptoms of infection at the time of inclusion in the study.
* Use of current antibiotic treatment or in the 2 weeks prior to inclusion in the study.
* Patients with malformations in the urinary tract
* Immunocompromised patients, diagnosed with cancer or AIDS.
* Urological cancer patients
* Patients who require continuous urine drainage (in the case of patients in the study arm) or hourly urine output measurement.
* Catheter insertion requiring more than one attempt.
* Inability to read and understand Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient experience for both types of catheterization | Through study completion, an average of 9 months
  For data collection, the technique of discussion groups will be used using a semi-structured script, which will serve for the identification of preferences and needs in daily life and for training and information for the use of the devices of catheterised patients. The discussion groups will be audio-recorded, transcribed and moderated by a researcher with experience in this field who does not have a therapeutic relationship with the participants.
Self-perceived general health status using 5 dimensions of 5 levels each, and a VAS ranging from 0 to 100. | Day 28 after inclusion
  The following instrument is administered to participants: EuroQol-5 Dimensions-5 Levels. A questionnaire that measures the patient's health status from a physical, psychological and social point of view. It consists of the descriptive system EQ-5D, which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels ranging from no problems to extreme problems. This decision results in a 1-digit number for each dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. In addition, it also features the EQ Visual Analogue Scale (EQ VAS), which records the patient's self-rated health on a visual analogue scale, where the endpoints are labelled "The best health you can imagine" (100) and "The worst health you can imagine" (0). The VAS can be used as a quantitative measure of health outcomes that reflect the patient's own judgement.
Quantitively assessed self-perceived catheter-related experience | Day 28 after inclusion
  Rethink Medical developed a specific instrument created in the context of this project based on the experience of our previous studies. The questionnaire aims to assess the self-perceived quality of life of catheterised patients and includes 29 questions that collect data on the prescription of the bladder catheter and on the accessories used (collection bag, cap or others), questions related to acceptability, usability and satisfaction in relation to the catheter and the accessories used, adverse events and changes in habits associated with the catheterisation and emotions perceived at the beginning and during the use of the bladder catheter. In order to quantitatively assess the answers, the statements will include multiple answer options, single options and answers with scores on a scale of 1 to 10.

SECONDARY OUTCOMES:
Rate and magnitude of infections (symptomatic and asymptomatic) | Day 28 after inclusion
  The number of urinary tract infections will be obtained from the analysis of urine samples taken from patients. The research staff will take two samples from each patient, one at the time of inclusion in the study and another at the follow-up visit, four weeks after the insertion of the probe, coinciding with the change of the catheter. The presence of pathogenic microorganisms in quantities greater than or equal to 1,000 CFU/ml will determine the presence of infection, while, in the absence of symptoms of infection, a determination of microorganisms greater than or equal to 100,000 CFU/ml will indicate asymptomatic infection.
Catheter tip-positive culture rate | Day 28 after inclusion
  A 1 cm catheter between the fixation balloon of the bladder catheter will be sectioned in a sterile manner, sent in a sterile container to the microbiology laboratory to analyze and identify the type of microorganisms.
Number of adverse events related to catheterization | Day 28 after inclusion
  The type and number of adverse events will be recorded: accidental disconnection of the catheter, obstruction, pain, loss of urine per catheter, haematuria and accidental spills caused by the professional during the moment of insertion.
Indication of antibiotic treatments | Day 28 after inclusion
  The antibiotic that has been administered associated with the use of the catheter will be recorded.
Total costs of each type of catheterization (cost-effectiveness) per quality-adjusted life year (QALY) of catheterized participants | Through study completion, an average of 9 months
  The costs derived from the catheterization, such as the consumption of consumable materials and resources, diagnostic tests (urine cultures and catheter cultures and biofilm analysis) will be collected. The budgetary impact derived from the incorporation of T-Control® into the service portfolio of Spanish hospitals will be included. The main outcome measure will be the incremental cost per quality-adjusted life year (QALY) gained, a generic health measure that combines information on life expectancy with the patient's quality of life, the latter measured through the EuroQoL-5 Dimensions-5 Levels instrument. The perspective of the analysis will be that of the hospital, in which only direct healthcare costs will be included.
The workload perceived by health professionals participating in the study. | Through study completion, an average of 9 months
  The following instrument is administered to health professionals: National Aeronautics and Space Administration - Task Load Index. This questionnaire is a subjective, multidimensional evaluation tool that qualifies the perceived workload to evaluate the effectiveness of a task, system or equipment or other aspects of performance. The questionnaire evaluates 6 dimensions (mental, physical and temporal demand, performance, effort and frustration) allowing to rate them in a 1 (lowest) to 10 (highest) scale.
Opinion of healthcare professionals of the devices used during the study | Through study completion, an average of 9 months
  The following instrument is administered to health professionals: Health professional satisfaction questionnaire. A questionnaire specifically developed by Rethink Medical to quantitatively measure preferences, problems and advantages encountered with the devices used. This questionnaire includes a first section with 12 statements regarding the catheter insertion process, the health professionals will rate these statements for both devices used during the clinical trial in a 1 to 5 scale depending if they agree (5) or not (1) with the statements. The second section is intended for health professionals to make a comparison between both devices through 11 statements for which they will have to indicate which device best fits these statements according to their opinion, being able to choose only one device for each statement. Finally, the questionnaire consists of a free section in which health professionals can write any comments or suggestions).

CONTACTS AND LOCATIONS:
Overall Officials: José Medina-Polo, Dr., Principal Investigator — Hospital Universitario 12 de Octubre
Locations (2):
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife

IPD SHARING:
Plan to Share IPD: Yes
The requests for participant-level data and/or statistical code can be made in writing to info@rethinkmedical.es. The final trial dataset generated and/or analysed during the study may be available on reasonable request to the research coordinator and Sponsor.
Supporting Information: Study Protocol
Time Frame: Starting 2 months after publication.
Access Criteria: Review requests and criteria for reviewing requests will be carried out by the Principal Investigators and Sponsor.